CLINICAL TRIAL: NCT06789575
Title: Comparison of Bupivacaine Wound Infiltration Versus Wound Instillation to Minimize Postoperative Pain After Thyroid Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hussin Abd elhakim, residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Wound Infilt/InstThyroid Surg
Record Dates: First submitted 2025-01-18; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Surgery
MeSH Terms: interventions — Bupivacaine; Epinephrine; Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group S (Active Comparator): mixture will instilled over the incision before the closure of the incision the patients will receive the content of a syringe (10 ml of bupivacaine 0.25% , 15 μg adrenaline and 70 ml Lidocaine ).
  Interventions: Drug: Bupivacaine; Drug: Adrenaline; Drug: Lidocaine (drug)
- Group F (Active Comparator): will recieve the mixture by injection inside the wound before the closure of the incision the patients will receive the content of a syringe (10 ml of bupivacaine 0.25% , 15 μg adrenaline and 70 ml Lidocaine ).
  Interventions: Drug: Bupivacaine; Drug: Adrenaline; Drug: Lidocaine (drug)

INTERVENTIONS:
Drug: Bupivacaine — the patients will receive the content of a syringe (10 ml of bupivacaine 0.25%)
Drug: Adrenaline — the patients will receive the content of a syringe 15 μg adrenaline
Drug: Lidocaine (drug) — the patients will receive the content of a syringe 70 ml Lidocaine .

SUMMARY:
Pain management following thyroidectomies, which can cause mild to moderate postoperative pain, particularly in the first 24 hours following surgery, has received little attention . The incision of the wound, neck hyperextension, retraction of the wound margins during surgery, and dissection are the main reasons of post-thyroidectomy discomfort . After thyroid surgery, pain management improves patients' quality of life and facilitates a speedy return to regular daily activities.

the aim of the study to evaluate the effects of bupivacaine instillation after thyroidectomy against infiltration into the surgical field in order to reduce postoperative discomfort following thyroid surgery.

DETAILED DESCRIPTION:
Pain management following thyroidectomies, which can cause mild to moderate postoperative pain, particularly in the first 24 hours following surgery, has received little attention . The incision of the wound, neck hyperextension, retraction of the wound margins during surgery, and dissection are the main reasons of post-thyroidectomy discomfort . After thyroid surgery, pain management improves patients' quality of life and facilitates a speedy return to regular daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Normal thyroid function patients of both genders scheduled for thyroid surgery will included in this study
* If they are over the age of 18
* If they had an ASA score (American Society of Anesthesiology) I, II.
* A Score of Mallampati I , II.

Exclusion Criteria:

* Patient refused to participate in the study.
* Patients will be excluded if they have any analgesic medication or corticosteroid drug prior surgery or
* A known or suspected allergy to local anesthetics,
* if the duration of surgery is greater than 5 h and if a major complication of surgery or anesthesia (major bleeding, allergy to anesthetic products).
* Patients who have lateral neck dissection associated with Thyroid surgery are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Total analgesic consumption | 24 hours
  Total analgesic consumption at 1st. 24 hours postoperative

IPD SHARING:
Plan to Share IPD: Undecided